CLINICAL TRIAL: NCT00880490
Title: A Randomized, Double-blind, Five-period, Placebo and Active-controlled,Cross-over, Multi-centre, Study Evaluating Single Administration of Three Doses of Inhaled PT005 in Patients With Moderate-to-Severe COPD, Compared to Open- Label Marketed Formoterol (FORADIL® AEROLIZER®) as an Active Control
Brief Title: Study to Evaluate the Safety and Efficacy of Inhaled PT005 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Chief Medical Officer, Pearl Therapeutics, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT0050801
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Inhaled PT005 2.4 mcg
  Interventions: Drug: Inhaled PT005
- 2 (Experimental): Inhaled PT005 4.8 mcg
  Interventions: Drug: Inhaled PT005
- 3 (Experimental): Inhaled PT005 9.6 mcg
  Interventions: Drug: Inhaled PT005
- 4 (Placebo Comparator): Inhaled Placebo
  Interventions: Drug: Inhaled placebo
- 5 (Active Comparator): Formoterol Fumarate 12 mcg (Foradil Aerolizer)
  Interventions: Drug: Formoterol Fumarate 12 mcg (Foradil Aerolizer)

INTERVENTIONS:
Drug: Inhaled PT005 — single dose, inhaled
  Arms: 1
Drug: Inhaled PT005 — single dose, inhaled
  Arms: 2
Drug: Inhaled PT005 — single dose, inhaled
  Arms: 3
Drug: Inhaled placebo — single dose, inhaled
  Arms: 4
Drug: Formoterol Fumarate 12 mcg (Foradil Aerolizer) — single dose, Formoterol Fumarate 12 mcg administered via the Aerolizer
  Other Names: Foradil Aerolizer
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of inhaled PT005 compared to placebo and Formoterol Fumarate (Foradil Aerolizer) in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* 40 - 80 years of age
* Fluency in written and spoken English
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* A measured post-salbutamol FEV1/FVC ratio of < or = 0.70
* A measured post-salbutamol FEV1 > or = 40 and < or = 80% of predicted normal values
* Demonstrated reversibility to a short acting beta agonist by either >12% and >150 ml improvement in baseline FEV1, 30 minutes following administration of 4 puffs of salbutamol MDI or an absolute improvement of >200 ml in baseline FEV1, 30 minutes following administration of 4 puffs of salbutamol MDI.
* Competent at using the inhalation device

Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 24 weeks of Screening
* Poorly controlled COPD in prior 6-weeks, defined as the occurrence of acute worsening of COPD requiring corticosteroids or antibiotics or acute worsening of COPD requiring treatment prescribed by a physician
* Clinically significant medical conditions
* Lower respiratory tract infection requiring antibiotics in past 6 weeks
* Clinically significant abnormal ECG
* Clinically significant uncontrolled hypertension
* Positive Hepatitis B surface antigen or Hepatitis C antibody
* Cancer that has not been in complete remission for at least 5 years
* History of hypersensitivity to any beta2-agonists or any study drug component
* History of severe milk protein allergy
* Known or suspected history of alcohol or drug abuse
* Medically unable to withhold short acting bronchodilators for 8-hours
* Use of the medications below in specified time interval prior to Screening: 12-weeks: depot corticosteroids, intra-articular corticosteroids; 4 weeks: ICS >1000 μg/day of fluticasone propionate or equivalent, non-potassium sparing diuretics, P-glycoprotein inhibitors, CYP3A4 inhibitors; 1 week: tiotropium; 48 hours: oral beta agonists, long acting beta agonists, theophylline, zariflukast, montelukast, zileuton; 8 hours: ipratropium or ipratropium/salbutamol combination product, inhaled short acting beta agonists, xanthine containing foods
* Use of the following medications is prohibited: tricyclic antidepressants, monoamine oxidase (MAO) inhibitors, beta-adrenergic antagonists, anticonvulsants (barbiturates,hydantoins, and carbamazepine and phenothiazines
* Receiving long-term-oxygen or nocturnal oxygen therapy for >12 hours a day
* Diagnosis of sleep apnea that is uncontrolled
* Participation in acute phase of pulmonary rehabilitation in prior 4 weeks or will enter acute phase of pulmonary rehabilitation program during study
* Unable to comply with study procedures
* Affiliated with Investigator site
* Questionable validity of consent
* A positive drug of abuse test at Screening lives prior to Screening, whichever is longer

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in one second (FEV1) area under the curve from 0 to 12 hours [AUC(0-12)] from test day baseline across the three doses of inhaled PT005 compared with placebo. | Serial FEV1 measured over 12 hours

SECONDARY OUTCOMES:
Time to onset of action (>10% improvement in FEV1 from baseline) | Serial FEV1 measured over 12 hours
Peak FEV1 | Serial FEV1 measured over 12 hours
Trough FEV1 | Serial FEV1 measured over 12 hours
Peak inspiratory capacity (IC) | Serial IC measured over 12 hours
Peak expiratory flow rate (PEFR) | Serial PEFR measured over 12 hours
Forced vital capacity (FVC) | Serial FVC measured over 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, M.D., Study Director — Pearl Therapeutics, Inc.
Locations (5):
- Australia (3):
  - Woolcock Institute of Medical Research, Glebe, New South Wales
  - Australian Clinical Research Organisation, Auchenflower, Queensland
  - Mater Hospital, South Brisbane, Queensland
- New Zealand (2):
  - Primorus Clinical Trials, Christchurch
  - P3 Research, Wellington

REFERENCES:
- [Derived] Quinn D, Seale JP, Reisner C, Fischer T, Golden M, Fernandez C, Darken P, St Rose E, Thomas M, Tardie G, Orevillo C. A randomized study of formoterol fumarate in a porous particle metered-dose inhaler in patients with moderate-to-severe COPD. Respir Med. 2014 Sep;108(9):1327-35. doi: 10.1016/j.rmed.2014.06.009. Epub 2014 Jul 3. PMID 25060541